CLINICAL TRIAL: NCT01249391
Title: Splinting to Treat Interphalangeal Joint Deformity in Hand Osteoarthritis(Splint OA Study)
Brief Title: Splinting to Treat Hand Osteoarthritis
Acronym: SPLINTOA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Imperial College London, Imperial College London
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JROHH051
Record Dates: First submitted 2010-11-25; First posted 2010-11-29 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2011-07

CONDITIONS: Hand Osteoarthritis
Keywords: Hand; osteoarthritis; splint; pain; deformity; function
MeSH Terms: conditions — Osteoarthritis; Pain; Congenital Abnormalities | interventions — Splints

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (splinting) (Active Comparator): Splinting of nominated joint in this group
  Interventions: Device: Splinting
- Control (No Intervention): Observation and usual treatment only.

INTERVENTIONS:
Device: Splinting — Gutter thermoplastic custom-made splint for nominated joint, to be worn at night-time for consecutive nights for 3 months
  Arms: Intervention (splinting)

SUMMARY:
Osteoarthritis (OA) is the most common form of arthritis and the hand is the most frequently affected site.Interphalangeal (IP) joints (the small joints of the fingers) are often involved causing pain, progressive loss of hand function and deformity. Deviation, or bending to the side, of IP joints (IPJs) with significant functional and cosmetic consequences for the individual is common. There are no drugs which can slow the disease process so there is reliance on symptomatic treatment such as pain relief and hand therapy. Joint thermoplastic splinting (moulded plastic splints that are custom-made) is employed by hand therapists in other settings, but to the investigators knowledge no studies have formally investigated the effect of splinting in IP OA.

By resting inflamed tissues and correcting joint alignment, a beneficial role for splinting in IP OA is likely. In this study, the investigators want to test whether thermoplastic splinting of deviated IP joints due to OA will 1) improve joint alignment 2) ameliorate soft tissue inflammation, and whether as a consequence 3) pain and overall hand function will be improved.

Adults with hand OA with 'affected' IP joints (symptoms from OA associated with deviation of the joint on X-ray)will be recruited from a specialist hand osteoarthritis clinic. Initially this will be for distal IP (DIP) joints. In the intervention group (30 patients), an 'intervention' joint for splinting will be identified as the most painful deviated DIP joint in the past week leading up to enrolment. Up to 3 other 'affected' DIP joints on either hand will not be splinted but will be monitored as 'control' joints. In the control group (15 patients), an affected joint will be monitored but not splinted. Assessment of joint pain, hand function by a hand therapist, deformity (by X-ray)and joint inflammation will take place at baseline, during and at the end of splinting period of 3 months, and also at 6 months,to assess whether any changes are persistent. In this way, the efficacy of splinting of IP joints in OA will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 90
* Definite diagnosis of IPJ osteoarthritis (American College of Rheumatology criteria for OA)
* A previous radiograph of the hands with changes consistent with OA
* Either, Intervention group: At least 2 'affected' IPJs (symptomatic (>2/10 average pain on 0-10 scale in past week) and radiological OA associated with 10 degrees of either radial or ulnar deviation of the joint evident clinically and on Xray)
* OR Control group: At least 1 'affected' IPJ (symptomatic (>2/10 average pain on 0-10 scale in past week) and radiological OA associated with 10 degrees of either radial or ulnar deviation of the joint evident clinically and on X-ray)
* Stable oral therapy for month prior to study entry e.g. non steroidal anti-inflammatory drugs (NSAIDs)
* Capable of providing written informed consent

Exclusion Criteria:

* Contraindication to splinting e.g. allergy to materials
* Planned surgery during study period
* Oral, intramuscular or intraarticular steroids within 3 months of study entry
* Intraarticular hyaluronans to any nominated IP joints within 6 months of study entry
* Not resident in UK
* Pregnancy
* Other inflammatory arthritis
* History of psoriasis
* Participation in other intervention trials
* Patients with any uncontrolled or severe medical problems which in the opinion of the investigator makes them unsuitable for study participation
* Unable to give informed written consent in English

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pain in nominated joint | 3 months
  Assessed via numerical rating scale

SECONDARY OUTCOMES:
Radiological deviation of nominated joint | 3 months
  Degrees of radial or ulnar deviation of joint will be assessed radiographically.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Watt, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Watt FE, Kennedy DL, Carlisle KE, Freidin AJ, Szydlo RM, Honeyfield L, Satchithananda K, Vincent TL. Night-time immobilization of the distal interphalangeal joint reduces pain and extension deformity in hand osteoarthritis. Rheumatology (Oxford). 2014 Jun;53(6):1142-9. doi: 10.1093/rheumatology/ket455. Epub 2014 Feb 8. PMID 24509405